CLINICAL TRIAL: NCT04666389
Title: The Role of Statins in the Prevention of Contrast-induced Acute Kidney Injury in Patients With Cardiovascular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Olga Mironova, Associate Professor, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09/2020
Record Dates: First submitted 2020-12-01; First posted 2020-12-14 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Contrast-induced Acute Kidney Injury; Cardiovascular Diseases
Keywords: contrast-induced acute kidney injury; contrast-associated acute kidney injury; contrast media; cardiovascular diseases; computer tomography
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Placebo Comparator): No statins being used for prevention
  Interventions: Drug: Atorvastatin
- Low-dose statin therapy (Active Comparator): Atorvastatin 40 mg
  Interventions: Drug: Atorvastatin
- High-dose statin therapy (Active Comparator): Atorvastatin 80 mg
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — To compare the preventive role of low- and high-dose statin regimens in the prevention on contrast-induced acute kidney injury in statin-naive patients with cardiovascular diseases undergoing computer tomography with intravenous contrast media administration

SUMMARY:
The aim of the study is to assess the role of statins and different dosage regimens in the prevention of contrast-induced acute kidney injury in patients with cardiovascular diseases requiring intravenous contrast media administration before computer tomography

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Indications for computer tomography with intravenous contrast media administration
* Cardiovascular diseases (arterial hypertension, arrhythmia etc)

Exclusion Criteria:

* Pregnancy
* Statin therapy before inclusion in the study
* Acute coronary syndromes
* Contraindications for statins administration
* Patients with chronic kidney disease stages 4-5
* Contraindications for computer tomography with contrast media administration
* Nephrotoxic drugs use (NSAIDS, vancomycin etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Contrast-induced acute kidney injury | 48-72 hours after contrast media administration
  Contrast induced acute kidney injury is defined as the 25% rise (or 0,5 mg/dl) of serum creatinine from baseline assessed 48 hours after administration of contrast media.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Mironova, MD PhD, Principal Investigator — Sechenov University
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasin AA, Mironova OI, Fomin VV. [The atorvastatin effects on the prevention of contrast-induced acute kidney injury during computed tomography with contrast media]. Ter Arkh. 2022 Oct 24;94(9):1057-1061. doi: 10.26442/0403660.2022.09.201845. Russian. PMID 36286755
- See also: Vasin AA, Mironova OIu, Fomin VV. The atorvastatin effects on the prevention of contrast-induced acute kidney injury during computed tomography with contrast media. Terapevticheskii Arkhiv (Ter. Arkh.). 2022;94(9):1057-1061. — https://doi.org/10.38109/2225-1685-2022-3-84-88
- See also: Vasin A.A., Mironova O.I., Fomin V.V. Intravenous contrast induced acute kidney injury prevention with high doses of statins. Eurasian heart journal. 2022;(3):84-88. (In Russ.) — https://doi.org/10.38109/2225-1685-2022-3-84-88
- See also: Vasin AA, Mironova OIu, Fomin VV. Contrast-induced acute kidney injury after computed tomography with contrast media in patients with cardiovascular diseases. Consilium Medicum. 2021;23(12):928-930. — https://doi.org/10.26442/20751753.2021.12.201162